CLINICAL TRIAL: NCT01000155
Title: A Phase II Pharmacodynamic Investigation of the Efficacy of Vorinostat to Induce Fetal Hemoglobin in Adults With Severe Sickle Cell Disease Who Have Not Benefitted From Prior Therapy
Brief Title: Efficacy of Vorinostat to Induce Fetal Hemoglobin in Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study terminated early due to slow accrual.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Maureen Okam, MD, MPH, Associate Physician, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-237
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: fetal hemoglobin; vorinostat; HDAC inhibitor; SAHA
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat (Experimental): Patients received vorinostat in a pulsed fashion, once a day for 3 consecutive days every week to a maximum dose of 400 mg per dose (1200 mg/wk), for 12 to 16 weeks at the maximum dose. The first 3 patients were enrolled in an intrapatient dose escalation schedule of 100 mg/d, then 200 mg/d, each for 3 consecutive days a week for 4 weeks, and then 400 mg/d, 3 consecutive days per week for 16 weeks. The last 2 patients were enrolled to receive 400 mg/d, 3 consecutive days per week for 12 weeks, without an initial dose escalation.
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat
  Other Names: SAHA

SUMMARY:
Sickle Cell Disease (SCD) is a hereditary anemia that causes the red blood cells to change their shape from a round and doughnut-like shape to a half-moon/crescent, or sickled shape. People who have SCD have a different type of hemoglobin (protein that carries oxygen). This different type of hemoglobin makes the red blood cells change into a crescent shape under certain conditions. Sickle-shaped cells are a problem because they often get stuck in the blood vessels blocking the flow of blood and can cause inflammation and injury to important areas of the body. All babies are born with hemoglobin called fetal hemoglobin (HbF). Soon after birth, HbF production slows down and another hemoglobin called adult hemoglobin (HbA) is made. Clinical studies have shown that increasing the amount of HbF in the blood may prevent sickling of the red blood cells. Vorinostat has been used in the treatment of cancers and in other research studies and information from those suggests that it may help treat SCD by increasing the amount of HbF in the blood. The purpose of this research study is to determine the effectiveness and safety of vorinostat when used to treat SCD.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of vorinostat (suberoylanilide hydroxamic acid, SAHA), when administered orally, in a pulsed fashion, once-a-day for 3 consecutive days every week, in inducing a 4% absolute increase or a 100% increase in fetal hemoglobin percent levels (HbF%) in subjects with severe sickle cell disease who have failed prior therapy.
* To characterize the safety and tolerability.

Secondary

* To assess the effect of vorinostat on F-cell levels.
* To determine the changes in y-globin, B-globin and E-globin RNA levels during treatment with vorinostat.
* To describe the dose-response characteristics of vorinostat in inducing fetal hemoglobin in sickle cell disease.

Exploratory

* To determine the extent and duration of global histone acetylation with intermittent vorinostat dosing.
* To correlate the status of polymorphisms near the BCL11A, c-myb, and HBB gene loci, all of which are associated with levels of fetal hemoglobin, to assess for an association of polymorphism status with therapeutic response to vorinostat.
* To evaluate red blood cell rheology before and after treatment with vorinostat.

STATISTICAL DESIGN:

This was a single stage design to evaluate induction of HbF on treatment with target enrollment of 15 patients. A 25% success rate was considered evidence of activity in this patient population while 5% success rate deemed ineffective. If at least 3 patients achieved success, the treatment would be considered promising. With 15 eligible patients, the probability of observing this was 0.76 assuming a true rate of 25% and 0.04 assuming a true rate of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease
* Clinically significant disease defined as at least 1 painful episode per year averaged over the previous 3 years or a history of priapism, stroke, acute chest syndrome, avascular necrosis, multi-organ failure or the need for chronic narcotic medications for pain from sickle cell disease
* Must have failed a previous attempt at treatment with hydroxyurea defined as the inability to achieve a significant absolute increase in % fetal hemoglobin or the inability to tolerate hydroxyurea treatment due to severe side effects such as but not limited to myelosuppression, gastrointestinal symptoms, edema or hepatic enzyme elevations or have contraindications to hydroxyurea
* 18 years of age or older
* Hematologic laboratory values as outlined in the protocol
* Non-hematologic laboratory values as outlined in the protocol
* Must agree not to donate blood or other bodily fluid while taking the study drug and for 28 days thereafter
* Women of child-bearing potential (WCBP) must have a negative serum pregnancy test 72 hours or less prior to starting treatment
* Women of child-bearing potential and men must agree to use 2 forms of adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Subjects with hemoglobin SC or SB+ thalassemia
* Subjects on chronic transfusion program
* Subjects who have received RBC transfusions cannot have >15% adult hemoglobin
* Known positive status for HIV, active hepatitis B or hepatitis C
* Pregnant or breast feeding women
* Individuals with a history of malignancy are ineligible except for the following circumstances. Individuals with a history of malignancy are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancer are eligible if diagnosed and adequately treated within the past 5 years: cervical or breast cancer in situ, and basal cell or squamous cell carcinoma of the skin
* Subjects with a history of thrombosis or other reason (other than sickle cell disease) for enhanced thrombotic risk
* Subjects with unresolved infections
* Severe or uncontrolled medical conditions that could compromise study participation
* Subjects on fetal hemoglobin inducing agents
* Subjects on any other experimental treatment within 90 days of the first dose of study drug or who have not recovered from the side effects of such therapy
* Known allergic reaction to a histone deacetylase inhibitor
* Subjects who have received valproic acid for treatment of epilepsy within 30 days of enrollment
* Subjects who have received any HDAC inhibitors other than valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Okam, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vorinostat
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Arm/Group | Vorinostat
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 37 [21 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Fetal Hemoglobin (HbF%) Induction Success Rate
Description: Success will be defined by comparing the maximum HbF% on study drug to the HbF% at baseline. An absolute increase in HbF% of 4% of more, or an increase to 100% or more of baseline in patients with HbF under 4% at baseline will be considered a success. HbF% induction success rate is calculated as the count of successes divided by the count of patients in the analysis population.
Time Frame: HbF% was measured at baseline and weekly on treatment. Median duration of treatment was 3 months.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Vorinostat
Number analyzed (Participants) | 5
proportion of patients | 0.20 [.01 to .65]

2. Secondary Outcome: F-Cell Percentage Level
Description: F-cell percentage levels were estimated based on established methods.
Time Frame: Measured at baseline and end of treatment, up to 16 weeks.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (Full Range); unit: F-cell percentage
Arm/Group | Vorinostat
Number analyzed (Participants) | 5
F-cell percentage
  Baseline | 9.8 [NA to NA] — This information was not provided at the time of the analysis and the data are no longer accessible.
  End of Treatment | 12.1 [NA to NA] — This information was not provided at the time of the analysis and the data are no longer accessible.

3. Secondary Outcome: γ-globin to β-globin Ratio
Description: Levels of peripheral blood γ-globin to β-globin messenger RNA were estimated based on established methods. The ratio of γ-globin to β-globin was then calculated.
Time Frame: Measured at baseline and end of treatment, up to 16 weeks.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (Full Range); unit: Change in γ-globin to β-globin ratio
Arm/Group | Vorinostat
Number analyzed (Participants) | 5
Change in γ-globin to β-globin ratio | 0.89 [0.34 to 1.4]

ADVERSE EVENTS:
Time Frame: Assessed weekly throughout treatment from time of first dose and up to day 30 post-treatment. Median duration of treatment was 3 months.
Description: Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3. Maximum grade toxicity by type was calculated within each group.
Arm/Group | Vorinostat
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat (N=5)
Constitutional, other (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat (N=5)
Necrosis, pancreas (Gastrointestinal disorders) | 1
IV116 (Renal and urinary disorders) | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Stenosis (incl anastomotic) duodenum (Gastrointestinal disorders) | 1
Bilirubin (Investigations) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The trial did not meet it's accrual goal due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No